CLINICAL TRIAL: NCT03728127
Title: Effect of the Brazilian Cardioprotective Diet and Nuts on Cardiometabolic Parameters in Post-acute Myocardial Infarction: a Randomized Clinical Trial (DICA-NUTS Study)
Brief Title: Brazilian Cardioprotective Diet and Nuts in Post-acute Myocardial Infarction
Acronym: DICA-NUTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DICA-NUTS; U1111-1259-8105 (Other: Universal Trial Number - World Health Organization (UTN-WHO))
Record Dates: First submitted 2018-10-29; First posted 2018-11-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DicaBr group and nuts (DCBN) (Experimental): Brazilian cardioprotective diet plus 30g/day of mixed nuts (10g of peanuts, 10g of cashew nuts and 10g of Brazil nuts)
  Interventions: Dietary Supplement: Brazilian cardioprotective diet plus 30g/day of mixed nuts
- DicaBr group (DCB) (Active Comparator): Brazilian cardioprotective diet
  Interventions: Dietary Supplement: Brazilian cardioprotective diet

INTERVENTIONS:
Dietary Supplement: Brazilian cardioprotective diet — Brazilian cardioprotective diet prescription
  Arms: DicaBr group (DCB)
Dietary Supplement: Brazilian cardioprotective diet plus 30g/day of mixed nuts — Brazilian cardioprotective diet plus 30g/day of nuts (10g of peanuts, 10g of cashew nuts and 10g of Brazil nuts)
  Arms: DicaBr group and nuts (DCBN)

SUMMARY:
Coronary artery disease (CAD) is the leading cause of death worldwide. Dietary patterns and functional foods may play an important role in the management of cardiovascular risk factors such as overweight and dyslipidemia, as well as inflammation and oxidative stress. However, little is known regarding the effect of diets or specific nutrients on these parameters in individuals with acute myocardial infarction (AMI). The Brazilian Cardioprotective Diet (DicaBr) is based on Brazilian nutritional guidelines and also in a unique and ludic nutritional strategy. In a pilot study, this diet was effective in reducing blood pressure (intragroup comparison) and body weight (intergroup comparison) in individuals with established cardiovascular disease (CVD). However, the effectiveness of this dietary pattern supplemented with different kind of nuts is unknown. The aim of this study is to evaluate the effect of the DicaBr supplemented or not with 30g/day of different nuts on cardiometabolic parameters in patients with recent AMI. In this parallel randomized controlled trial, 388 patients ≥40 years with a recent diagnosis of AMI (60 to 180 days) will be allocated to one of two study groups: 1) DicaBr group (DCB, control group); or 2) DicaBr group supplemented with mixed nuts (DCBN, intervention group). All patients will receive the same dietary prescription, the DCBN group also will receive 30g/day of nuts (10g of peanuts, 10g of cashew nuts and 10g of Brazilian nuts). A pilot study including 100 individuals who will receive only peanuts (30g/day) will be conducted. The primary outcome will be LDL-cholesterol (LDL-c) levels after 16 weeks. In the baseline and at the end of the study (16 weeks), lipid and glycemic profile and anthropometric indexes will be evaluated in both groups; inflammatory and oxidative stress markers, and adipokines will be evaluated in a subsample. It is expected that DicaBr supplemented with nuts will be superior to DicaBr alone to benefit patients with AMI regarding cardiometabolic parameters.

ELIGIBILITY:
Inclusion Criteria: Patients ≥ 40 years with previous AMI (60 to 180 days).

Exclusion Criteria:

* Clinical indication of myocardial revascularization surgery (graf /bypass);
* HIV positive in treatment/AIDS;
* Chronic inflammatory diseases;
* Cancer;
* Chemical dependency/alcoholism;
* Chronic use of anti-inflammatories, anticonvulsants and immunosuppressive drugs;
* Pregnancy or lactation;
* Wheelchair users without conditions of anthropometric evaluation;
* Extreme obesity (BMI ≥40kg / m²);
* Use of dietary supplements;
* Rejection/allergy to oilseed consumption;
* Participation in other randomized studies at the time of enrollment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
LDL-c | Changes in LDL-c after 16 weeks
  Low-density lipoprotein cholesterol (LDL-c), in mg/dL: LDL-c will be detected by Martins´mathematical formula

SECONDARY OUTCOMES:
TC | Changes in TC after 16 weeks
  Total cholesterol (TC), in mg/dL
HDL-c | Changes in HDL-c after 16 weeks
  High-density lipoprotein cholesterol (HDL-c), in mg/dL
TG | Changes in TG after 16 weeks
  Serum triglycerides (TG), in mg/dL
VLDL-c | Changes in VLDL after 16 weeks
  Very low-density lipoprotein cholesterol (VLDL-c), in mg/dL; serum triglycerides, (in mg/dL) divided by 5 will be used to report VLDL-c in mg/dL
NHDL-c | Changes in NHDL-c after 16 weeks
  Non-HDL cholesterol (NHDL-c), in md/dL; total cholesterol (in mg/dL) and high-density lipoprotein cholesterol (in mg/dL) will be combined to report NHDL-c in mg/dL
TG/HDL-c | Changes in TG/HDL-c after 16 weeks
  TG/HDL-c ratio (TG/HDL-c), in mg/dL; serum triglycerides (in mg/dL) and high-density lipoprotein cholesterol (in mg/dL) will be combined to report TG/HDL-c in mg/dL
Castelli I index | Changes in Castelli I index after 16 weeks
  TC/HDL-c ratio, in mg/dL; total cholesterol (in mg/dL) and high-density lipoprotein cholesterol (in mg/dL) will be combined to report Castelli I index in mg/dL
Castelli II index | Changes in Castelli II index after 16 weeks
  LDL-c/HDL-c ratio, in mg/dL; low-density lipoprotein cholesterol (in mg/dL) and high-density lipoprotein cholesterol (in mg/dL) will be combined to report Castelli II index in mg/dL
FG | Changes in FG after 16 weeks
  Fasting glucose (FG), in mg/dL
INS | Changes in INS after 16 weeks
  Serum insulin (INS), in mU/L
HbA1C | Changes in HbA1C after 16 weeks
  glycated hemoglobin (HbA1C), in %
HOMA-IR | Changes in HOMA-IR after 16 weeks
  Homeostasis model assessment-insulin resistance, defined according to: [FG (in mmol) x INS (in UI/mL) ÷ 22.5]
BW | Changes in BW after 16 weeks
  Body weight, in kg
BMI | Changes in BMI after 16 weeks
  Body mass index (BMI), in kg/m^2; weight (in kg) and height (in meters) will be combined to report BMI in kg/m^2
WC | Changes in WC after 16 weeks
  Waist circumference (WC), in cm
HC | Changes in HC after 16 weeks
  Hip circumference, in cm
WHR | Changes in WHR after 16 weeks
  Waist-to-hip ratio (WHR); waist circumference (in cm) and hip circumference (in cm) will be combined to report WHR
WHt | Changes in WHt after 16 weeks
  Waist-to-height ratio (WHt); waist circumference (in cm) and height (in meters) will be combined to report WtH, in cm/m

CONTACTS AND LOCATIONS:
Overall Officials: Aline Marcadenti, PhD, Principal Investigator — Hospital do Coracao; Alexandre Cavalcanti, PhD, Study Director — Hospital do Coracao; Bernardete Weber, PhD, Study Chair — Hospital do Coracao; Angela Bersh-Ferreira, PhD, Study Chair — Hospital do Coracao; Enilda Lara, PhD, Study Chair — Hospital do Coracao; Rachel Machado, MSc, Study Chair — Hospital do Coracao; Lucas Ribeiro, RD, Study Chair — Hospital do Coracao
Locations (9):
- Brazil (9):
  - Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte
  - Instituto de Cardiologia/Fundação Universitária de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas da Universidade Federal do Paraná (HC-UFPR), Curitiba
  - Hospital de Clínicas da Universidade Federal de Goiás (HC-UFG), Goiânia
  - Universidade Federal de Alagoas (UFAL), Maceió
  - Hospital de Clínicas de Porto Alegre - Universidade Federal do Rio Grande do Sul (HCPA-UFRGS), Porto Alegre
  - Instituto Nacional de Cardiologia (INC), Rio de Janeiro
  - Universidade Federal do Maranhão (UFMA), São Luís
  - Hospital do Coração (HCor), São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Data and materials will be available upon reasonable request for the corresponding author, after filling a specific form provided by IP-HCor and considering institutional data sharing politics.
Supporting Information: Study Protocol
Time Frame: Data will be available after the main paper publication.
Access Criteria: Link for design paper (study protocol):
  https://pubmed.ncbi.nlm.nih.gov/34470656/

REFERENCES:
- [Derived] Bersch-Ferreira AC, Weschenfelder C, Vieira Machado RH, Nakagawa Santos RH, Riley TM, da Silva LR, Miyada DHK, Sady ERR, de Abreu-Silva EO, Laranjeira LN, de Quadros AS, Dos Santos JL, Souza GC, Parahiba SM, Fayh APT, Bezerra DS, Carvalho APPF, Machado MMA, Vasconcelos SML, Santos MVR, de Figueiredo Neto JA, Dias LPP, Zaina Nagano FE, de Almeida CCP, Moreira ASB, de Oliveira RD, Rogero MM, Sampaio GR, da Silva Torres EAF, Weber B, Cavalcanti AB, Marcadenti A. Effects of mixed nuts as part of a Brazilian Cardioprotective diet on LDL-cholesterol in adult patients after myocardial infarction: a multicenter randomized controlled clinical trial. Nutr J. 2024 Oct 1;23(1):118. doi: 10.1186/s12937-024-01020-5. PMID 39354558
- [Derived] Marcadenti A, Weber B, Bersch-Ferreira AC, Machado RHV, Torreglosa CR, de Sousa Lara EM, da Silva LR, Santos RHN, Miyada DHK, Sady ERR, Costa RP, Piegas L, de Abreu-Silva EO, de Quadros AS, Weschenfelder C, Dos Santos JL, Souza GC, Parahiba SM, Fayh APT, Bezerra DS, Carvalho APPF, Machado MMA, Vasconcelos SML, Araujo J, de Figueiredo Neto JA, Dias LPP, Nagano FEZ, de Almeida CCP, Moreira ASB, Gapanowicz DP, Purgatto E, Rogero MM, Sampaio GR, da Silva Torres EAF, Duarte GBS, Cavalcanti AB. Effects of a Brazilian cardioprotective diet and nuts on cardiometabolic parameters after myocardial infarction: study protocol for a randomized controlled clinical trial. Trials. 2021 Sep 1;22(1):582. doi: 10.1186/s13063-021-05494-0. PMID 34470656